CLINICAL TRIAL: NCT04808479
Title: FOA Title: HEAL Initiative: Behavioral Research to Improve MAT: Behavioral and Social Interventions to Improve Adherence to Medication-Assisted Treatment for Opioid Use Disorders (R61/R33 Clinical Trial Optional
Brief Title: Effectiveness of a CBT-based mHealth Intervention Targeting MOUD Retention, Adherence, and Opioid Use
Acronym: UCimFREE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC imFREE phase1&RCT
Record Dates: First submitted 2021-02-08; First posted 2021-03-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC imFREE Smartphone application intervention (Experimental): The imFREE condition is a 32-week tailored, interactive text messaging intervention targeting buprenorphine treatment retention and adherence as well as opioid use and associated health consequences. Following a face-to-face CBT session with a clinician, participants receive CBT skills training via daily text messaging, with content themes around relapse prevention, adherence behaviors, and personalized plans to overcome risk factors for treatment discontinuation.
  Interventions: Behavioral: imFREE mCBT
- Health Education and pamphlet (Active Comparator): The mHealth condition will provide participants with a manualized health psychoeducation session of equivalent duration to the face-to-face CBT session delivered to imFREE participants. Content focuses on various dimensions of health and well-being. Subsequent to this session participants will receive an informational pamphlet regarding BUP and the importance of adherence. the mHealth component of the intervention comprises text reminders for scheduled MM appointments.
  Interventions: Behavioral: mHealth ED

INTERVENTIONS:
Behavioral: imFREE mCBT — The imFREE condition is a 32-week tailored, interactive text messaging intervention targeting buprenorphine treatment retention and adherence as well as opioid use and associated health consequences. Following a face-to-face CBT session with a clinician, participants receive CBT skills training via daily text messaging, with content themes around relapse prevention, adherence behaviors, and personalized plans to overcome risk factors for treatment discontinuation.
  Other Names: imFREE
  Arms: UC imFREE Smartphone application intervention
Behavioral: mHealth ED — The mHealth condition will provide participants with a manualized health psychoeducation session of equivalent duration to the face-to-face CBT session delivered to imFREE participants. Content focuses on various dimensions of health and well-being. Subsequent to this session participants will receive an informational pamphlet regarding BUP and the importance of adherence. the mHealth component of the intervention comprises text reminders for scheduled MM appointments.
  Other Names: Manualized Health Psychoeducation
  Arms: Health Education and pamphlet

SUMMARY:
The focus of this study is to examine the effectiveness of imFREE relative to mHealth ED in facilitating treatment retention and adherence and reducing opioid use among adults with OUD initiating BUP treatment.

There are two specific aims: (1) to test the effectiveness of imFREE, delivered in conjunction with medical management with buprenorphine (imFREE + MM), relative to mHealth ED + MM, in facilitating buprenorphine treatment retention and adherence in a population of individuals with OUD initiating MM (N=200). (2) To evaluate the cost-effectiveness of imFREE.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* DSM-5 diagnosis of OUD
* no more than 2 weeks from the date of BUP induction
* able to read and comprehend English at the 6th grade level (determined by REALM)
* able to provide informed consent
* presently owns a mobile phone that can send and receive text messages

EXCLUSION CRITERIA

Participants must not have:

1. Life threatening or unstable medical illness requiring treatment or making participation difficult
2. Dependence on alcohol or other illicit substances for which medical detoxification is imminently needed
3. Presence of acute psychiatric symptoms warranting intensive treatment or hospitalization (e.g., acute suicidality or mania).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence self-report form. Unannounced medication count by phone | Monthly from date of randomization, for up to 6 months, or until study completion, whichever comes first.
  Self-report of Treatment adherence to buprenorphine collected in self-report forms. Unannounced medication count by phone. Research staff will call participants and ask them to count out the remaining buprenorphine films left in their prescription.

SECONDARY OUTCOMES:
DSM-V Checklist | Baseline
  Assessing the presence of opiate use disorder

OTHER OUTCOMES:
European Addiction Severity Index | Baseline, month 3, month 6
  The Addiction Severity Index is a relatively brief, semi-structured interview designed to provide important information about aspects of a client's life that may contribute to his/her substance abuse syndrome.Assessment of addiction severity and frequency of alcohol/drug use.
Urine drug screen | Throughout six months, monthly
  Confirming absence/presence of opiates and buprenorphine
Medical Management (MM) attendance | Throughout six months, monthly
  Retention in buprenorphine treatment my reviewing number of MM sessions attended

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Tarzana Treatment Center, Tarzana, California, United States